CLINICAL TRIAL: NCT04456283
Title: Prospective Analysis of the Survival of Patients With a Reduction in the Number of Lymph Nodes in Rectal Cancer After Neoadjuvant Chemoradiotherapy
Brief Title: Survival of Patients With a Reduction in the Number of Lymph Nodes in Rectal Cancer After Neoadjuvant Chemoradiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: SERGIO CARLOS NAHAS (Unknown); CAIO SERGIO NAHAS (Unknown); Ivan Cecconello (Unknown); Ulysses Ribeiro Junior (Unknown)
Responsible Party: Principal Investigator, Leonardo Alfonso Bustamante, Post doctoral fellow, University of Sao Paulo
Other Study IDs: 9076078
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cancer of Rectum; Lymph Node Disease
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Incomplete pathological response with less than 12 LN.: Patients with incomplete pathological response after Chemoradiation theraphy for Rectal Cancer and less than 12 lymph nodes
  Interventions: Behavioral: Survival
- Incomplete pathological response with 12 or more LN.: Patients with incomplete pathological response after Chemoradiation theraphy for Rectal Cancer and 12 lymph or more nodes
  Interventions: Behavioral: Survival
- Complete pathological response with less than 12 LN.: Patients with complete pathological response after Chemoradiation theraphy for Rectal Cancer and less than 12 lymph nodes
  Interventions: Behavioral: Survival
- Complete pathological response with 12 or more LN.: Patients with complete pathological response after Chemoradiation theraphy for Rectal Cancer and 12 lymph or more nodes
  Interventions: Behavioral: Survival

INTERVENTIONS:
Behavioral: Survival — 5 year survival after Chemoradiation theraphy for Rectal Cancer

SUMMARY:
Objective: To analyze the survival of patients with a reduction in the number of resected LN in patients submitted to neoadjuvant and total excision of the mesorectum with rectal cancer.

Expected results:

Survival rate between patients Complete Pathologic Response with less than 12 LN and 12 or more LN.

To determine the difference in survival between patients with less than 12 LN in complete versus incomplete response.

DETAILED DESCRIPTION:
According to the International Union Against Cancer a minimum of 12 lymph nodes (LN) should be obtained in the surgical specimen for colorectal cancer staging. Recent studies have reported that the use of neoadjuvant chemoradiotherapy (QRN) may result in failure to obtain the minimum number of LN in the piece in 30-52% of patients. Objective: To analyze the survival of patients with a reduction in the number of resected LN in patients submitted to neoadjuvant and total excision of the mesorectum with rectal cancer. Patients and methods: From January 2013 to January 2015, patients with rectal cancer were submitted to QRN (5-FU and 5040 Gys) followed by total excision of mesorectum with ligation of the inferior mesenteric vessels in their roots. Patients with T3, T4 and / or N + staging that were up to 10 cm from the anal border were included. Patients whose treatment with neoadjuvant chemoradiotherapy was incomplete or who had significant delays in re- staging and / or performing the surgery were excluded. All were staged by rectal examination, colonoscopy, chest and abdominal CT, and pelvic MRI, and also re-staged 8 weeks after neoadjuvant termination, operated and submitted to total excision of the mesorectum. The patients were divided into 4 groups: a) Incomplete pathological response with less than 12 LN. b) Incomplete pathological response with 12 or more LN. c) Complete pathological response with less than 12 LN. d) Complete pathological response with 12 or more LN. The possible variables related to the number of LN obtained and related to general and disease free survival were studied.

Expected results:

To analyze the survival rate between patients Complete Pathologic Response with less than 12 LN and 12 or more LN. To determine the difference in survival between patients with less than 12 LN in complete versus incomplete response. Demonstrate that patients with complete pathologic response and less than 12 LN have a disease-free survival equal to or better than patients with 12 LN or more.

ELIGIBILITY:
Inclusion Criteria: Patients with a biopsy-proven mid and low rectal adenocarcinoma located within 10 cm from the anal verge, stage cT3-4N0M0 or cT (any)N + M0, and patients with low (< 5 cm from anal verge) cT2N0 of distal rectum because of the risk of needing an abdominoperineal resection.

-

Exclusion Criteria: Patients with synchronous colorectal cancer or other non-colorectal cancers, stage IV disease, rectal cancer in the setting of inflammatory bowel disease or familial adenomatous polyposis, palliative resections, previous pelvic radiotherapy, significant comorbidities that prevent curative surgical resection and/or CRT, concurrent participation in another research protocol involving therapeutic intervention

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with mid and low rectal cancer within 10 cm from the anal verge, stage cT3-4N0M0 or cT (any)N + M0
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
5 years Survival | 5 years
  5 years Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine School, Sao Paulo University, São Paulo, Brazil